CLINICAL TRIAL: NCT06223269
Title: A Phase III Open-Label, Multicenter, Randomized, Controlled Clinical Trial to Evaluate the Safety and Efficacy of realSKIN® to Provide Complete Wound Closure of Mixed-Depth, Full-Thickness Burn Wounds as an Alternative to Autografting
Brief Title: Safety and Efficacy of realSKIN® to Provide Complete Wound Closure of Burn Wounds as an Alternative to Autografting
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: XenoTherapeutics, Inc. (Other)
Collaborators: Joseph M. Still Research Foundation, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: realSKIN-003
Record Dates: First submitted 2023-06-15; First posted 2024-01-25 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Burns Degree Third; Burn (Disorder); Burn Degree Second; Thermal Burn; Wound Heal
Keywords: Full-thickness Burn; Complete Wound Closure; Durable Wound Closure; Autograft Alternative; 3rd Degree Burn; Mixed-Depth Burn; Partial-thickness Burn; 4th Degree Burn; Xenotransplant; Xenograft; Skin Xenotransplant; realSKIN
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: Open-label, interventional, controlled, randomized, multicenter clinical trial. Each patient represents both the experimental and control group, to be evaluated in isolated but comparable settings. The use of an intra-patient comparator allows for a matched control to eliminate significant underlying differences. Treatment assignment will be randomized to receive either realSKIN or a surgically harvested autograft.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Skin Xenotransplant (Experimental): After surgical preparation of the wound beds, subjects will receive approximately 100 square centimeters of realSKIN® at one site, and autograft at the other site, per the standard of care, in accordance with the randomization schedule.
  Interventions: Drug: Skin Xenotransplant
- Autograft (Active Comparator): The comparator control for the study is autografting: the current standard of care procedure for the treatment of severe burns involves the removal of a sheet of healthy skin from an uninjured site on the patient and using it to cover the original burn wound to achieve complete and durable wound closure.
  Interventions: Procedure: Autograft(ing)

INTERVENTIONS:
Drug: Skin Xenotransplant — realSKIN® is a live biotherapeutic, bi-layered, split-thickness, membranous, skin xenotransplant wound dressing manufactured from living porcine skin sourced from genetically engineered, alpha-1,3-galactosyltransferase knock-out (GalT-KO) porcine (Sus scrofa) donors under aseptic conditions.
  realSKIN® is topically applied to a surgically prepared wound bed via sutures or staples and may be trimmed to fit the shape and size of the wound area.
  Other Names: realSKIN®
  Arms: Skin Xenotransplant
Procedure: Autograft(ing) — Autograft(ing) is the current standard of care procedure for the treatment of severe burns. The procedure involves the removal of a sheet of healthy skin, i.e. autologous (self) skin harvesting, from an uninjured site on the patient and using it to cover the original burn wound.
  Arms: Autograft

SUMMARY:
To evaluate the safety and efficacy of realSKIN® to provide complete wound closure of mixed-depth, full-thickness burn wounds as an alternative treatment to autografting.

DETAILED DESCRIPTION:
This study is a Phase 3 open-label, interventional, controlled, randomized, multicenter clinical trial. It is comprised of an estimated 50 men and women aged 18 years and older who experienced severe and extensive, mixed-depth and full-thickness thermal burn wounds up to 50% TBSA requiring surgical excision and skin grafting for which autografting is clinically indicated.

The comparator control for the study is autografting, the current standard of care procedure for the treatment of severe burns, which involves the removal of healthy skin from an uninjured site on the patient and using it to cover the original burn wound to achieve complete and durable wound closure.

After surgical preparation of the wound bed, subjects will receive approximately 100 square centimeters of realSKIN at a predesignated wound site and separately, autografting at an alternate site, per the standard of care, in accordance with the randomization schedule.

Thus, each patient represents both the experimental and control group, to be evaluated in isolated but comparable settings. The use of an intra-patient comparator allows for a matched control to eliminate significant underlying differences, including immunologic, physiologic, and scarring variable inherent in this patient population that may impact wound healing at the treatment sites.

After surgical excision to remove nonviable tissue or previously applied temporary wound dressings, two wound treatment sites of comparable area and depth will be identified.

Treatment assignment will be randomized to receive either realSKIN or a surgically harvested autograft. The pre-identified treatment sites must each be a wound area of comparable depth that is not contiguous (e.g., "sharing a common border or touching") to ensure the interpretability of the efficacy results.

Additionally, two unaffected areas of the patient's intact, healthy skin will be prospectively identified to provide sources of autografts for the control site and realSKIN treatment site (e.g., patient skin harvest sites.) These pre-identified regions may be in the same anatomic area or from two separate but comparable areas, depending on the amount of intact native patient skin available.

ELIGIBILITY:
Inclusion Criteria:

1. The subject, or the subject's legally authorized representative (LAR), provides written informed consent to participate in this study
2. Males or females age greater than or equal to 18 years old
3. Total Burn Surface Area (TBSA) <50% to include mixed depth and full-thickness burn wounds as defined as "primarily full-thickness (FT) and deep-partial (DPT) thermal burns (e.g. >60% of the total burn area should be FT and DPT) before debridement", and full-thickness burns for which surgical intervention is clinically indicated
4. Having a mixed depth thermal burn wound including full thickness requiring skin grafting
5. Biological females must have a negative serum pregnancy test at Screening and must not be nursing
6. All subjects must agree to use a protocol-approved method of contraception for a minimum of 3 months following realSKIN placement, which includes a barrier method plus one or more of the following:

   * Hormonal contraceptives (e.g., birth control pills, skin patches, vaginal rings, and the Depo-Provera shot)
   * Intrauterine device (IUD)
   * Male or female condoms with spermicide
   * Diaphragm with spermicide
   * Permanent tubal occlusive birth control system
7. Sufficient area of burn wound for realSKIN and comparator autograft placement to not be located on face or hands or having a target graft site centered on high-impact areas such as joints, weight-bearing areas (e.g. soles of feet), or the inguinal region, per Investigator's judgment

Exclusion Criteria:

1. Pregnant or lactating women
2. Documented history of infection with human immunodeficiency virus (HIV) or other condition(s) that in the opinion of the Investigator may compromise patient safety or study objectives
3. Immunosuppressive medication regimens e.g. antineoplastics, high dose steroids (>10 mg prednisone/day), TNF alpha inhibitors, calcineurin inhibitors (cyclosporine, tacrolimus), anti- proliferative agents, and other immunomodulators
4. Active malignancy, including those requiring surgery, chemotherapy, and/or radiation in the past 5 years; non-metastatic basal or squamous cell carcinoma of the skin and cervical carcinoma in situ are allowed
5. Use of any experimental or investigational drugs within 30 days prior to placement of realSKIN
6. Previously received a porcine or other xenogeneic tissue product, including but not limited to: glutaraldehyde fixed porcine or bovine bioprosthetic heart valve replacements and glutaraldehyde fixed porcine dermal matrix (e.g., EZ Derm)
7. Patients with advanced or unstable/uncontrolled comorbid conditions, such as advanced renal disease, diabetes mellitus and liver disease
8. Patients with HbA1c ≥ 10.0%; specimen must be obtained for screening purposes if current (within past 3 months) value is not available
9. Patients with a history of chronic end stage renal disease defined as MDRD CrCL < 15mL/min or receiving chronic dialysis
10. Patients with a history of chronic liver disease or cirrhosis (Child-Pugh Score C); evidence of acute or chronic hepatitis B infection based on documented HBV serology testing
11. Known documented history of Hepatitis B, Hepatitis C, Treponema pallidum, Cytomegalovirus, herpes or varicella zoster; note: Successfully treated hepatitis C patients without evidence of end stage liver disease is allowed; if HCV antibody reactive, then HCV RNA must be undetectable
12. Recent (within 3 months prior to study enrollment) MI, unstable angina leading to hospitalization, uncontrolled, CABG, PCI, carotid surgery or stenting, cerebrovascular accident, transient ischemic attack, endovascular procedure, or surgical intervention for peripheral vascular disease or plans to undergo a major surgical or interventional procedure (e.g., PCI, CABG, carotid or peripheral revascularization)
13. Presence of venous or arterial vascular disorder directly affecting the area of burn wound
14. Pre-existing haemolytic anemia
15. Chronic malnourishment as determined by Investigator
16. Inhalation injury as determined by bronchoscopic exam if available, or diagnosis at the time of screening
17. Systemic anticoagulation at the time of treatment or INR > 2
18. Documented evidence of wound infection at Screening
19. Evidence of sepsis at Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Complete Wound Closure at Post-Treatment Day 28 (± 7 days) | Post-Treatment Day 28 (± 7 days)
  Complete wound closure is defined as >95% skin re-epithelization in an area of the treatment site without drainage or dressing requirements by Post-Treatment Day 28 (± 7 days).
  Durable wound closure is defined as confirmation of complete wound closure in an area of the treatment site at two consecutive evaluations, spaced by no less than 14 days and no more than 5 months.
  Post-Treatment is defined as time elapsed following autografting and treatment with realSKIN, and is not necessarily time elapsed from time of initial time of injury (i.e. in cases where an interim wound dressings were employed prior to autografting.)
Percent Area of Treatment Sites Autografted | Post-Treatment Month 4 (± 1 month)
  Percent area of treatment sites autografted is the sum of the percent areas at each assessment/visit.

SECONDARY OUTCOMES:
Pain at the Patient Skin Harvest Sites | Post-Treatment Month 4 (± 1 month)
  Visual Analogue Scale (VAS) scale range from 0 (no pain) to 10 (worst pain). Pain scores assessed up to Post-Treatment Month 4 (± 1 month) are averaged for the summary statistics.
Exploratory Endpoint: Evaluate realSKIN treatment sites for the existence of residual porcine cell populations at Post-Treatment Month 4 (± 1 month). | Post-Treatment Month 4 (± 1 month)
  3 mm skin biopsies will be obtained from enrolled and treated patients of this study who volunteer to provide samples for analysis at post-treatment Month 4 (± 1 month).

CONTACTS AND LOCATIONS:
Overall Officials: Bounthavy Homsombath, MD, Principal Investigator — JMS BURN CENTER AT DOCTORS HOSPITAL OF AUGUSTA
Locations (4):
- United States (4):
  - Arizona Burn Center Valleywise Health, Phoenix, Arizona
  - JMS Burn Center at Doctors Hospital, Augusta, Georgia
  - MaineHealth Maine Medical Center, Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibson ALF, Holmes JH 4th, Shupp JW, Smith D, Joe V, Carson J, Litt J, Kahn S, Short T, Cancio L, Rizzo J, Carter JE, Foster K, Lokuta MA, Comer AR, Smiell JM, Allen-Hoffmann BL. A phase 3, open-label, controlled, randomized, multicenter trial evaluating the efficacy and safety of StrataGraft(R) construct in patients with deep partial-thickness thermal burns. Burns. 2021 Aug;47(5):1024-1037. doi: 10.1016/j.burns.2021.04.021. Epub 2021 Apr 23. PMID 34099322
- [Background] Albritton A, Leonard DA, Leto Barone A, Keegan J, Mallard C, Sachs DH, Kurtz JM, Cetrulo CL Jr. Lack of cross-sensitization between alpha-1,3-galactosyltransferase knockout porcine and allogeneic skin grafts permits serial grafting. Transplantation. 2014 Jun 27;97(12):1209-15. doi: 10.1097/TP.0000000000000093. PMID 24798308
- [Background] Bruccoleri RE, Matthew MK, Schulz JT. Methods in obtaining split-thickness skin grafts from skin reduction surgery specimens. Springerplus. 2016 May 25;5(1):690. doi: 10.1186/s40064-016-2330-2. eCollection 2016. PMID 27350924
- [Background] Burd A, Chiu T. Allogenic skin in the treatment of burns. Clin Dermatol. 2005 Jul-Aug;23(4):376-87. doi: 10.1016/j.clindermatol.2004.07.019. PMID 16023933
- [Background] Denner J. Paving the Path toward Porcine Organs for Transplantation. N Engl J Med. 2017 Nov 9;377(19):1891-1893. doi: 10.1056/NEJMcibr1710853. No abstract available. PMID 29117497
- [Background] Deschamps JY, Roux FA, Sai P, Gouin E. History of xenotransplantation. Xenotransplantation. 2005 Mar;12(2):91-109. doi: 10.1111/j.1399-3089.2004.00199.x. PMID 15693840
- [Background] Ericsson TA, Takeuchi Y, Templin C, Quinn G, Farhadian SF, Wood JC, Oldmixon BA, Suling KM, Ishii JK, Kitagawa Y, Miyazawa T, Salomon DR, Weiss RA, Patience C. Identification of receptors for pig endogenous retrovirus. Proc Natl Acad Sci U S A. 2003 May 27;100(11):6759-64. doi: 10.1073/pnas.1138025100. Epub 2003 May 9. PMID 12740431
- [Background] Fishman JA, Scobie L, Takeuchi Y. Xenotransplantation-associated infectious risk: a WHO consultation. Xenotransplantation. 2012 Mar-Apr;19(2):72-81. doi: 10.1111/j.1399-3089.2012.00693.x. PMID 22497509
- [Background] Godehardt AW, Rodrigues Costa M, Tonjes RR. Review on porcine endogenous retrovirus detection assays--impact on quality and safety of xenotransplants. Xenotransplantation. 2015 Mar-Apr;22(2):95-101. doi: 10.1111/xen.12154. Epub 2015 Jan 31. PMID 25641488
- [Background] Johnson RM, Richard R. Partial-thickness burns: identification and management. Adv Skin Wound Care. 2003 Jul-Aug;16(4):178-87; quiz 188-9. doi: 10.1097/00129334-200307000-00010. PMID 12897674
- [Background] Kitala D, Kawecki M, Klama-Baryla A, Labus W, Kraut M, Glik J, Ryszkiel I, Kawecki MP, Nowak M. Allogeneic vs. Autologous Skin Grafts in the Therapy of Patients with Burn Injuries: A Restrospective, Open-label Clinical Study with Pair Matching. Adv Clin Exp Med. 2016 Sep-Oct;25(5):923-929. doi: 10.17219/acem/61961. PMID 28028957
- [Background] Leonard DA, Mallard C, Albritton A, Torabi R, Mastroianni M, Sachs DH, Kurtz JM, Cetrulo CL Jr. Skin grafts from genetically modified alpha-1,3-galactosyltransferase knockout miniature swine: A functional equivalent to allografts. Burns. 2017 Dec;43(8):1717-1724. doi: 10.1016/j.burns.2017.04.026. Epub 2017 Jun 8. PMID 28602591
- [Background] Leto Barone AA, Mastroianni M, Farkash EA, Mallard C, Albritton A, Torabi R, Leonard DA, Kurtz JM, Sachs DH, Cetrulo CL Jr. Genetically modified porcine split-thickness skin grafts as an alternative to allograft for provision of temporary wound coverage: preliminary characterization. Burns. 2015 May;41(3):565-74. doi: 10.1016/j.burns.2014.09.003. Epub 2014 Oct 16. PMID 25406888
- [Background] Martin SI, Wilkinson R, Fishman JA. Genomic presence of recombinant porcine endogenous retrovirus in transmitting miniature swine. Virol J. 2006 Nov 2;3:91. doi: 10.1186/1743-422X-3-91. PMID 17081300
- [Background] Meije Y, Tonjes RR, Fishman JA. Retroviral restriction factors and infectious risk in xenotransplantation. Am J Transplant. 2010 Jul;10(7):1511-6. doi: 10.1111/j.1600-6143.2010.03146.x. PMID 20642677
- [Background] Morozov VA, Wynyard S, Matsumoto S, Abalovich A, Denner J, Elliott R. No PERV transmission during a clinical trial of pig islet cell transplantation. Virus Res. 2017 Jan 2;227:34-40. doi: 10.1016/j.virusres.2016.08.012. Epub 2016 Sep 24. PMID 27677465
- [Background] Paradis K, Langford G, Long Z, Heneine W, Sandstrom P, Switzer WM, Chapman LE, Lockey C, Onions D, Otto E. Search for cross-species transmission of porcine endogenous retrovirus in patients treated with living pig tissue. The XEN 111 Study Group. Science. 1999 Aug 20;285(5431):1236-41. doi: 10.1126/science.285.5431.1236. PMID 10455044
- [Background] Patience C, Takeuchi Y, Weiss RA. Infection of human cells by an endogenous retrovirus of pigs. Nat Med. 1997 Mar;3(3):282-6. doi: 10.1038/nm0397-282. PMID 9055854
- [Background] Sen CK, Gordillo GM, Roy S, Kirsner R, Lambert L, Hunt TK, Gottrup F, Gurtner GC, Longaker MT. Human skin wounds: a major and snowballing threat to public health and the economy. Wound Repair Regen. 2009 Nov-Dec;17(6):763-71. doi: 10.1111/j.1524-475X.2009.00543.x. PMID 19903300
- [Background] Sheridan RL, Tompkins RG. Skin substitutes in burns. Burns. 1999 Mar;25(2):97-103. doi: 10.1016/s0305-4179(98)00176-4. No abstract available. PMID 10208382
- [Background] Shi M, Wang X, Okamoto M, Takao S, Baba M. Inhibition of porcine endogenous retrovirus (PERV) replication by HIV-1 gene expression inhibitors. Antiviral Res. 2009 Aug;83(2):201-4. doi: 10.1016/j.antiviral.2009.04.011. Epub 2009 May 3. PMID 19414036
- [Background] Weiner J, Yamada K, Ishikawa Y, Moran S, Etter J, Shimizu A, Smith RN, Sachs DH. Prolonged survival of GalT-KO swine skin on baboons. Xenotransplantation. 2010 Mar-Apr;17(2):147-52. doi: 10.1111/j.1399-3089.2010.00576.x. PMID 20522247
- [Background] Wilhelm M, Fishman JA, Pontikis R, Aubertin AM, Wilhelm FX. Susceptibility of recombinant porcine endogenous retrovirus reverse transcriptase to nucleoside and non-nucleoside inhibitors. Cell Mol Life Sci. 2002 Dec;59(12):2184-90. doi: 10.1007/s000180200017. PMID 12568344
- [Background] Wood JC, Quinn G, Suling KM, Oldmixon BA, Van Tine BA, Cina R, Arn S, Huang CA, Scobie L, Onions DE, Sachs DH, Schuurman HJ, Fishman JA, Patience C. Identification of exogenous forms of human-tropic porcine endogenous retrovirus in miniature Swine. J Virol. 2004 Mar;78(5):2494-501. doi: 10.1128/jvi.78.5.2494-2501.2004. PMID 14963150
- [Background] Wynyard S, Nathu D, Garkavenko O, Denner J, Elliott R. Microbiological safety of the first clinical pig islet xenotransplantation trial in New Zealand. Xenotransplantation. 2014 Jul-Aug;21(4):309-23. doi: 10.1111/xen.12102. Epub 2014 May 7. PMID 24801820
- [Background] Yue S, Zhang Y, Gao Y. A study on the susceptibility of allogeneic human hepatocytes to porcine endogenous retrovirus. Eur Rev Med Pharmacol Sci. 2015 Sep;19(18):3486-91. PMID 26439047
- [Background] Holzer PW, Leonard DA, Shanmugarajah K, Moulton KN, Ng ZY, Cetrulo CL Jr, Sachs DH. A Comparative Examination of the Clinical Outcome and Histological Appearance of Cryopreserved and Fresh Split-Thickness Skin Grafts. J Burn Care Res. 2017 Jan/Feb;38(1):e55-e61. doi: 10.1097/BCR.0000000000000431. PMID 27606556
- [Derived] Wu D, Zhao XS, Zhao HF, Xie JH, Wei HJ, Zhu NW. New Hope for the Treatment of Severe Skin Injury: Genetically Engineered Porcine Skin Xenotransplantation. Xenotransplantation. 2025 May-Jun;32(3):e70057. doi: 10.1111/xen.70057. PMID 40407357